CLINICAL TRIAL: NCT03122483
Title: Use of Blood Biomarkers and Biomarker Index to Aid in the Diagnosis of Obstructive Sleep Apnea (OSA)
Status: Completed | Type: Observational
Sponsor: Beckman Coulter, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SAB-03-15
Record Dates: First submitted 2017-04-17; First posted 2017-04-20 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- OSA: Blood biomarker results in subjects with obstructive sleep apnea.
  Interventions: Diagnostic Test: blood biomarker
- Non-OSA: Blood biomarker results in subjects without obstructive sleep apnea
  Interventions: Diagnostic Test: blood biomarker

INTERVENTIONS:
Diagnostic Test: blood biomarker

SUMMARY:
This multicenter prospective trial will evaluate the association between obstructive sleep apnea (OSA) and blood biomarkers in a representative population of consecutively enrolled symptomatic patients with a clinical suspicion of OSA.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent
* Male
* 18-70 years old
* Presentation with symptoms suggestive of obstructive sleep apnea
* Diagnostic sleep study
* Blood draw

Exclusion Criteria:

* Prior (within past year) or current therapy for sleep apnea
* Use of opioid pain medication, steroids or allopurinol (within past 30 days)
* Use of chronic anti-inflammatory drugs (within past 7 days)
* Active cancer under current treatment or monitoring

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Symptomatic patients with a clinical suspicion of obstructive sleep apnea
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2017-07-14 (Actual)

PRIMARY OUTCOMES:
Identification of OSA in high-risk individuals | 1 day
  Identification of OSA in high-risk individuals

CONTACTS AND LOCATIONS:
Overall Officials: Paula C Southwick, PhD, Study Director — Beckman Coulter, Inc.
Locations (3):
- United States (3):
  - Sleep Center Orange County, Irvine, California
  - Brigham and Women's Hospital, Boston, Massachusetts
  - SleepMed, Columbia, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fleming WE, Ferouz-Colborn A, Samoszuk MK, Azad A, Lu J, Riley JS, Cruz AB, Podolak S, Clark DJ, Bray KR, Southwick PC. Blood biomarkers of endocrine, immune, inflammatory, and metabolic systems in obstructive sleep apnea. Clin Biochem. 2016 Aug;49(12):854-61. doi: 10.1016/j.clinbiochem.2016.05.005. Epub 2016 May 13. PMID 27184708